CLINICAL TRIAL: NCT02496221
Title: A Randomized, Double-blind, Single-dose, Placebo Controlled, 2-way Cross-over Study Evaluating Effect of Albiglutide on Cholecystokinin-induced Gallbladder Emptying in Fasting Healthy Subjects
Brief Title: A Study Evaluating the Effect of Albiglutide on Gallbladder Emptying in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201834
Record Dates: First submitted 2015-05-18; First posted 2015-07-14 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Cholecystokinin; ultrasonography; Albiglutide; Gallbladder ejection fraction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein; Sincalide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Albiglutide / Placebo or Placebo / Albiglutide (Experimental): In treatment period 1, subjects will receive Albiglutide 50 mg or Placebo subcutaneously (SC) after fasting overnight for at least 10 hours according to randomization schedule on Day 1. Subject will also receive CCK (Kinevac) infusion intravenously for a period of 50 minutes after fasting overnight for at least 10 hours on Day 4. After washout period of a minimum of 42 days in treatment period 2, subjects will receive same treatment according to randomization schedule in a cross-over fashion
  Interventions: Drug: Albiglutide 50 mg; Drug: Placebo; Drug: CCK (Kinevac)

INTERVENTIONS:
Drug: Albiglutide 50 mg — Albiglutide 50 mg pen is a single-use fixed dose, fully disposable pen injector system for SC delivery in the abdomen containing 67 mg lyophilized albiglutide and 0.65 mL diluents designed to deliver a dose of 50 mg in a volume of 0.5 mL after reconstitution
Drug: Placebo — Placebo is a single-use fixed dose, fully disposable pen injector system for SC delivery of 0.5 mL injector volume in the abdomen
Drug: CCK (Kinevac) — CCK (Kinevac) will be infused intravenously. Kinevac is supplied in vials containing 5 microgram (mcg)/vial. Infusion prepared aseptically by adding 5 mL of Sterile Water for Injection United States Pharmacopeia (USP) to the vial to create a solution of 1 mcg/mL. Infuse 0.003 mcg/kg dose in 100 mL of Sodium Chloride Injection USP, 0.9%

SUMMARY:
Albiglutide, a novel analogue of glucagon-like peptide-1 (GLP-1), has been developed and approved for the treatment of type 2 diabetes mellitus. The primary objective of this study is to assess if a single dose of albiglutide can affect cholecystokinin-induced gallbladder emptying. To make this assessment, each study participant will receive a dose of albiglutide and a dose of placebo followed by cholecystokinin (CCK) infusion and ultrasound measurement of the gallbladder.

The study will be comprised of two periods and 20 subjects. The screening visit will occur within 42 days of the start of Treatment Period 1. The Treatment Periods will be separated by a washout period of a minimum of 42 days. Subjects will return for a follow-up visit after 28 days following the last dose of albiglutide or placebo. The total duration of a subject's participation from Screening to Follow-up will be approximately 17.5 weeks.

This study is a post marketing commitment to the United States Food and Drug Administration (USFDA).

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age
* Healthy
* Have venous access sufficient to allow for intravenous (IV) infusion and blood sampling as per protocol
* Subject's body mass index (BMI) is >=18 kilogram (kg)/meter(m)^2 and <=30 kg/m^2
* Male or
* Female: if she is not pregnant (as confirmed by a test at screening and at other timepoints), not lactating, and at least one of the following conditions applies: a) cannot bear children OR b) agrees to follow contraception requirements defined in the protocol
* Capable of giving signed informed consent

Exclusion Criteria:

* Alanine aminotransferase (ALT) >1.5x Upper limit of normal (ULN)
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) > 450 milliseconds (msec)
* Systolic blood pressure is >=140 millimetre (mm) mercury (Hg) at Screening
* Diastolic blood pressure is >=90 mm Hg at Screening
* Heart rate is >100 beats/min at Screening
* Fasting triglyceride level >300 milligram/decilitre at Screening
* History of cholecystitis or other gallbladder disease
* History of gallstones, biliary motility dysfunction, or any condition rendering the subject unsuitable for ultrasonography assessments
* Prior cholecystectomy or any other gallbladder or biliary ducts procedure, prior ileal or gastric surgery, or any other medical procedure that precluded gallbladder emptying
* History of significant cardiovascular or pulmonary dysfunction prior to screening
* History of thyroid dysfunction
* History of intestinal obstruction, ileus, lap-band, gastrointestinal surgery or any other procedures that in the opinion of the investigator could influence gastric emptying (e.g., gastrectomy, gastric bypass)
* History of acute or chronic pancreatitis
* History of abdominal pain of unknown cause
* History of severe gastrointestinal disease, including gastroparesis, inflammatory bowel disease, Crohn's disease, or irritable bowel syndrome
* Personal or family history of multiple endocrine neoplasia type 2
* Personal or family history of medullary carcinoma of the thyroid
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days
* Current or past use of medications that may have significantly affected gastrointestinal and/or gallbladder motility or pancreatic or hepatobiliary systems
* History of regular alcohol consumption within 6 months of the study
* Urinary cotinine levels indicative of smoking or history of regular use of tobacco- or nicotine-containing products within 3 months prior to screening
* Subject has a history of significant weight loss or is currently attempting weight loss
* History of sensitivity or contraindication to any of the study medications or components thereof or a history of drug or other allergy
* Subject has previously received any GLP-1 mimetic compound (e.g., exenatide, liraglutide, lixisenatide, dulaglutide)
* A biliary pathology as assessed by ultrasound
* An abnormal (i.e., outside the normal reference range) thyroid function test assessed by thyroid stimulating hormone at screening
* An abnormal amylase or lipase test at screening
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result
* A positive pre-study drug/alcohol screen
* A positive test for Human immunodeficiency virus (HIV) antibody
* A screening ultrasound which demonstrates inadequate imaging of gallbladder, main pancreatic duct, or common duct
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56-day period
* The subject participated in a clinical trial and received an investigational product within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2015-10-13 (Actual); Study Completion 2015-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Shaddinger BC, Young MA, Billiard J, Collins DA, Hussaini A, Nino A. Effect of Albiglutide on Cholecystokinin-Induced Gallbladder Emptying in Healthy Individuals: A Randomized Crossover Study. J Clin Pharmacol. 2017 Oct;57(10):1322-1329. doi: 10.1002/jcph.940. Epub 2017 May 19. PMID 28543352
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 201834 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201834 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 201834 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201834 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201834 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201834 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201834 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were randomized to one of the two treatments in Treatment Period 1 followed by a wash-out period and crossed over to other treatment in Treatment Period 2.
Groups:
- Albiglutide 50 mg Followed by Placebo: Participants received Albiglutide 50 milligrams (mg) in Treatment Period 1 and Placebo in Treatment Period 2, each administered subcutaneously as a single dose, using a fully disposable pen injector system. Participants also received an intravenous infusion of cholecystokinin (sincalide) in each period.
- Placebo Followed by Albiglutide 50 mg: Participants received Placebo in Treatment Period 1 and Albiglutide 50 mg in Treatment Period 2, each administered subcutaneously as a single dose, using a fully disposable pen injector system. Participants also received an intravenous infusion of cholecystokinin (sincalide) in each period.
Period: Treatment Period 1 - 4 Days
Arm/Group | Albiglutide 50 mg Followed by Placebo | Placebo Followed by Albiglutide 50 mg
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Treatment Period 2 - 4 Days
Arm/Group | Albiglutide 50 mg Followed by Placebo | Placebo Followed by Albiglutide 50 mg
Started | 10 | 10
Completed | 8 | 9
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Albiglutide 50 mg and Placebo: In a total of two treatment periods, participants received Albiglutide 50 mg (A) and Placebo (P) (in a sequence of either A-P or P-A), each administered subcutaneously as a single dose, using a fully disposable pen injector system. Participants also received an intravenous infusion of cholecystokinin (sincalide) in each period.
Arm/Group | Albiglutide 50 mg and Placebo
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.8 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 15
  White - White/Caucasian/European Heritage | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Absolute Value of Gallbladder Ejection Fraction (Emax GEF) During Cholecystokinin (CCK) Infusion, as a Measure of Maximum Effect
Description: Gallbladder ejection fraction (EF) is defined as the reduction in gallbladder volume at any time point from Baseline divided by baseline gallbladder volume and multiplied by 100. Baseline gallbladder volume is the average of the 3 gallbladder volume measurements prior to CCK infusion on Day 4, for each treatment period. Gallbladder ultrasonography was done at Day 1 (-15, -10, and -5 minutes [min] relative to start of albiglutide/placebo injection) and Day 4 ([prior to CCK infusion] -15, -10, -5 min, followed by [during CCK infusion] every 5 min between 0 and 50 min, then [after CCK infusion] at 60, 70, and 80 min, relative to the start of CCK infusion). Adjusted mean and its standard error have been presented.
Time Frame: Day 4 in each treatment period
Population: Evaluable Subjects: Participants in the 'All Subjects' population who had gallbladder ultrasonography assessment pre-treatment and post-Baseline (during CCK infusion) for both periods. 'All Subjects' population comprised participants who received at least one dose of Investigational product.
Measure: Least Squares Mean (Standard Error); unit: Percent of gallbladder EF
Groups:
- Placebo: In one of the two treatment periods, participants received Placebo as a single subcutaneous dose, using a fully disposable pen injector system. Participants also received an intravenous infusion of cholecystokinin (sincalide) in this period.
- Albiglutide 50 mg: In one of the two treatment periods, participants received Albiglutide 50 mg as a single subcutaneous dose, using a fully disposable pen injector system. Participants also received an intravenous infusion of cholecystokinin (sincalide) in this period.
Arm/Group | Placebo | Albiglutide 50 mg
Number analyzed (Participants) | 17 | 17
Percent of gallbladder EF | 47.4352 (4.00997) | 38.4331 (4.00997)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide 50 mg; Test type: Superiority or Other; p = 0.1229, Mixed Models Analysis; Treatment (albiglutide or placebo), and period as fixed effects and participant as random effect; Mean Difference (Final Values) = -9.0021, 95% CI 2-sided [-20.5781 to 2.5739]

2. Primary Outcome: Area Under the Effect Curve for Gallbladder Ejection Fraction (AUEC GEF)
Description: Gallbladder ultrasonography was done at Day 1 (-15, -10, and -5 minutes [min] relative to start of albiglutide/placebo injection) and Day 4 ([prior to CCK infusion] -15, -10, -5 min, followed by [during CCK infusion] every 5 min between 0 and 50 min, then [after CCK infusion] at 60, 70, and 80 min, relative to the start of CCK infusion). Adjusted mean and its standard error have been presented.
Time Frame: Day 4 in each treatment period
Population: Evaluable Subjects
Measure: Mean (Standard Error); unit: %*min
Arm/Group | Placebo | Albiglutide 50 mg
Number analyzed (Participants) | 17 | 17
%*min | 1004.2510 (247.34751) | 458.2926 (247.34751)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide 50 mg; Test type: Superiority or Other; p = 0.1291, Mixed Models Analysis; Mean Difference (Final Values) = -545.9585, 95% CI 2-sided [-1260.00 to 168.0858]

3. Primary Outcome: Time at Which the Maximum Effect (Emax GEF) Occurred (TEMAXEF) During the CCK Infusion
Description: Gallbladder ultrasonography was done at Day 1 (-15, -10, and -5 minutes [min] relative to start of albiglutide/placebo injection) and Day 4 ([prior to CCK infusion] -15, -10, -5 min, followed by [during CCK infusion] every 5 min between 0 and 50 min, then [after CCK infusion] at 60, 70, and 80 min, relative to the start of CCK infusion).
Time Frame: Day 4 in each treatment period
Population: Evaluable Subjects
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | Albiglutide 50 mg
Number analyzed (Participants) | 17 | 17
Minutes | 37.64706 (13.1241) | 32.94118 (14.5836)

4. Primary Outcome: Maximum Gallbladder Ejection Fraction Value During CCK Infusion
Description: as for outcome 3
Time Frame: Day 1 and Day 4 in each treatment period
Population: Evaluable Subjects
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Albiglutide 50 mg
Number analyzed (Participants) | 17 | 17
Percentage | 44.5989 (5.11879) | 28.2997 (5.11879)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide 50 mg; Test type: Superiority or Other; p = 0.0317, Mixed Models Analysis; Treatment (albiglutide or placebo), and period as fixed effects and participant as random effect; Mean Difference (Final Values) = -16.2992, 95% CI 2-sided [-31.0762 to -1.5223]

5. Primary Outcome: Area Under the Effect Curve for Gallbladder Volume (AUEC VL)
Description: Gallbladder ultrasonography was done at Day 1 (-15, -10, and -5 minutes [min] relative to start of albiglutide/placebo injection) and Day 4 ([prior to CCK infusion] -15, -10, -5 min, followed by [during CCK infusion] every 5 min between 0 and 50 min, then [after CCK infusion] at 60, 70, and 80 min, relative to the start of CCK infusion). Adjusted mean and its standard error is presented.
Time Frame: Day 4 in each treatment period
Population: Evaluable Subjects
Measure: Mean (Standard Error); unit: mL*min
Arm/Group | Placebo | Albiglutide 50 mg
Number analyzed (Participants) | 17 | 17
mL*min | 610.5642 (91.00301) | 863.1741 (91.00301)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide 50 mg; Test type: Superiority or Other; p = 0.0291, Mixed Models Analysis; Treatment (albiglutide or placebo), and period as fixed effects and participant as random effect; Mean Difference (Final Values) = 252.6099, 95% CI 2-sided [29.5081 to 475.7117]

6. Primary Outcome: Maximum Absolute Change From Baseline in Value of Gallbladder Volume (Emax VL) During CCK Infusion, as a Measure of Maximum Effect
Description: Gallbladder ultrasonography was done at Day 1 (-15, -10, and -5 minutes [min] relative to start of albiglutide/placebo injection) and Day 4 ([prior to CCK infusion] -15, -10, -5 min, followed by [during CCK infusion] every 5 min between 0 and 50 min, then [after CCK infusion] at 60, 70, and 80 min, relative to the start of CCK infusion). Baseline gallbladder volume is the average of the 3 gallbladder volume measurements prior to CCK infusion on Day 4, for each treatment period. Adjusted mean and its standard error are presented.
Time Frame: Day 4 in each treatment period
Population: Evaluable Subjects
Measure: Mean (Standard Error); unit: Millilitre (mL)
Arm/Group | Placebo | Albiglutide 50 mg
Number analyzed (Participants) | 17 | 17
Millilitre (mL) | 8.8385 (1.39713) | 8.4637 (1.39713)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide 50 mg; Test type: Superiority or Other; p = 0.7961, Mixed Models Analysis; Treatment (albiglutide or placebo), and period as fixed effects and participant as random effect; Mean Difference (Final Values) = -0.3748, 95% CI 2-sided [-3.4109 to 2.6614]

7. Primary Outcome: Time at Which the Maximum Effect (Emax VL) Occurred (TEmax VL) During the CCK Infusion
Description: as for outcome 3
Time Frame: Day 4 in each treatment period
Population: Evaluable Subjects
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | Albiglutide 50 mg
Number analyzed (Participants) | 17 | 17
Minutes | 37.64706 (13.1241) | 32.94118 (14.5836)

8. Primary Outcome: Maximum Change From Baseline in Main Pancreatic Duct Diameter During CCK Infusion
Description: Pancreatic duct ultrasonography was done at Day 1 (-15, -10, and -5 minutes [min] relative to start of albiglutide/placebo injection) and Day 4 ([prior to CCK infusion] -15, -10, -5 min, followed by [during CCK infusion] every 5 min between 0 and 50 min, then [after CCK infusion] at 60, 70, and 80 min, relative to the start of CCK infusion). Baseline is the average of the three diameter assessments at -15, -10, and -5 minutes relative to start of CCK infusion on Day 4. Change from Baseline was calculated as the value at the indicated time point minus the Baseline value. Adjusted mean and its standard error are presented. Baseline was calculated as the value at the indicated time point minus the Baseline value. Only those participants available at the indicated time points were analyzed.
Time Frame: Day 4 in each treatment period
Population: Evaluable for Pancreatic: Participants with Baseline and post-Baseline pancreatic duct diameter values for both periods
Measure: Mean (Standard Error); unit: Centimetre (CM)
Arm/Group | Placebo | Albiglutide 50 mg
Number analyzed (Participants) | 6 | 5
Centimetre (CM) | 0.04359 (0.01373) | 0.04511 (0.01471)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide 50 mg; Test type: Superiority or Other; p = 0.9424, Mixed Models Analysis; Treatment (albiglutide or placebo), and period as fixed effects and participant as random effect; Mean Difference (Final Values) = 0.001526, 95% CI 2-sided [-0.045665 to 0.048717]

9. Primary Outcome: Maximum Change From Baseline in Common Bile Duct Diameter During CCK Infusion
Description: Common bile duct ultrasonography was done at Day 1 (-15, -10, and -5 minutes [min] relative to start of albiglutide/placebo injection) and Day 4 ([prior to CCK infusion] -15, -10, -5 min, followed by [during CCK infusion] every 5 min between 0 and 50 min, then [after CCK infusion] at 60, 70, and 80 min, relative to the start of CCK infusion). Baseline is the average of the three diameter assessments at -15, -10, and -5 minutes relative to start of CCK infusion on Day 4. Change from Baseline was calculated as the value at the indicated time point minus the Baseline value. Adjusted mean and its standard error have been presented.
Time Frame: Day 4 in each treatment period
Population: Evaluable for Bile: Participants with Baseline and post-Baseline common bile duct diameter values for both periods
Measure: Mean (Standard Error); unit: Centimetre (cm)
Arm/Group | Placebo | Albiglutide 50 mg
Number analyzed (Participants) | 17 | 17
Centimetre (cm) | 0.08814 (0.008308) | 0.07358 (0.008308)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide 50 mg; Test type: Superiority or Other; p = 0.0733, Mixed Models Analysis; Treatment (albiglutide or placebo), and period as fixed effects and participant as random effect; Mean Difference (Final Values) = -0.01456, 95% CI 2-sided [-0.030666 to 0.001554]

10. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Baseline is defined as Day 1 (pre-dose) visit. SBP and DBP were measured in a semi-supine position after 5 minutes of rest, at each indicated time point. Assessments were performed on Day -1, Day 1 (pre-dose), Day 2, Day 3 and 15 minutes (-15 min) prior to dosing and 80 min post dosing on Day 4. Change from Baseline was calculated as value at indicated time point minus Baseline value. Only those participants available at the indicated time points (represented by n=X,X in the category titles) were analyzed.
Time Frame: Day -1, Baseline Day 1(Pre-dose), Day 2, Day 3, and 15 minutes (-15 min) prior to dosing and 80 min post dosing on Day 4 in each treatment period and Follow-up (assessed up to a total of approximately 12 weeks)
Population: All Subjects
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | Albiglutide 50 mg
Number analyzed (Participants) | 18 | 20
Millimeters of mercury (mmHg)
  SBP, Period 1, Day 2, n=10, 10 | 2.5 (8.55) | 2.5 (8.29)
  SBP, Period 1, Day 3, n=10, 10 | 4.2 (6.86) | 4.3 (8.79)
  SBP, Period 1, Day 4 (-15 min), n=10, 10 | 4.8 (11.29) | 0.4 (10.16)
  SBP, Period 1, Day 4 (80 min), n=10, 10 | 2.2 (8.53) | 9.4 (7.23)
  SBP, Period 2, Day 2, n=8, 10 | 2.1 (9.70) | 0.0 (9.48)
  SBP, Period 2, Day 3, n=8, 10 | -2.5 (7.67) | -0.4 (8.63)
  SBP, Period 2, Day 4 (-15 min), n=8, 10 | 4.5 (9.15) | 0.8 (6.01)
  SBP, Period 2, Day 4 (80 min), n=8, 9 | 8.9 (9.63) | 4.7 (8.62)
  DBP, Period 1, Day 2, n=10, 10 | 2.9 (6.08) | -0.4 (9.22)
  DBP, Period 1, Day 3, n=10, 10 | 1.7 (5.25) | 3.2 (9.61)
  DBP, Period 1, Day 4 (-15 min), n=10, 10 | 6.3 (8.26) | 5.2 (8.63)
  DBP, Period 1, Day 4 (80 min), n=10, 10 | 2.2 (5.12) | 9.5 (6.65)
  DBP, Period 2, Day 2, n=8, 10 | -2.1 (8.37) | -4.3 (7.12)
  DBP, Period 2, Day 3, n=8, 10 | -3.4 (8.09) | -3.0 (10.15)
  DBP, Period 2, Day 4 (-15 min), n=8, 10 | 3.3 (5.23) | 0.0 (7.07)
  DBP, Period 2, Day 4 (80 min), n=8, 9 | 6.4 (6.30) | 0.4 (7.62)

11. Secondary Outcome: Change From Baseline in Heart Rate
Description: Baseline is defined as Day 1 (pre-dose) visit. Heart rate was measured in a semi-supine position after 5 minutes of rest, at each indicated time point. Assessments were performed on Day -1, Day 2, Day 3 and 15 minutes (-15 min) prior to dosing and 80 min post dosing on Day 4. Change from Baseline was calculated as value at indicated time point minus Baseline value. Only those participants available at the indicated time points (represented by n=X,X in the category titles) were analyzed.
Time Frame: Day -1, Baseline Day 1(Pre-dose), Day 2, Day 3, and 15 minutes (-15 min) prior to dosing and 80 min post dosing on Day 4 in each treatment period and Follow-up (a total of approximately 12 weeks)
Population: All Subjects
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Placebo | Albiglutide 50 mg
Number analyzed (Participants) | 18 | 20
Beats per minute (bpm)
  Period 1, Day 2, n=10, 10 | 2.4 (2.67) | 4.3 (4.60)
  Period 1, Day 3, n=10, 10 | 4.7 (6.72) | 7.9 (4.41)
  Period 1, Day 4 (-15 min), n=10, 10 | 3.8 (9.15) | 8.5 (4.74)
  Period 1, Day 4 (80 min), n=10, 10 | 1.4 (5.50) | 9.4 (7.59)
  Period 2, Day 2, n=8, 10 | 2.5 (7.91) | 4.2 (6.18)
  Period 2, Day 3, n=8, 10 | 3.4 (6.05) | 9.4 (8.19)
  Period 2, Day 4 (-15 min), n=8, 10 | 1.0 (2.78) | 6.3 (5.70)
  Period 2, Day 4 (80 min), n=8, 9 | 1.8 (3.58) | 6.3 (11.48)

12. Secondary Outcome: Number of Participants With Clinical Chemistry and Hematology Abnormalities of Potential Clinical Importance
Description: The following parameters were measured through blood sampling. Hematology: Hematocrit, Hemoglobin, Lymphocytes, Neutrophil Count, Platelet Count, While Blood Cell Count (WBC); Clinical Chemistry: Albumin, Calcium, Creatinine, Glucose, Magnesium, Phosphorus, Potassium, Sodium, Total carbon dioxide; Liver Function Tests: Alanine transaminase (ALT), Aspartate transaminase, Alkaline Phosphatase, Total Bilirubin, Total Bilirubin + ALT. Values were considered to be of potential clinical importance if they had a 'low' or 'high' flag with respect to a pre-defined clinical concern range. Only participants starting each period (represented by n=X) with a particular treatment were analyzed. The follow-up time point is not restricted to a treatment or treatment period.
Time Frame: Day -1 in each treatment period and Follow-up (at approximately Week 12)
Population: All Subjects
Measure: Number; unit: Participants
Groups:
- Albiglutide 50 mg and Placebo: In a total of two treatment periods, participants received Albiglutide 50 mg (A) and Placebo (P) (in a sequence of either A-P or P-A), each administered subcutaneously as a single dose, using a fully disposable pen injector system. Participants also received an intravenous infusion of a cholecystokinin (sincalide) in each period.
Arm/Group | Albiglutide 50 mg and Placebo
Number analyzed (Participants) | 20
Participants
  Clinical Chemistry, Albiglutide Period 1, n=10 | 1
  Clinical Chemistry, Placebo Period 2, n=8 | 2
  Clinical Chemistry, Follow-up, n=17 | 1
  Hematology, Albiglutide Period 1, n=10 | 1
  Hematology, Albiglutide Period 2, n=10 | 1

13. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters
Description: Single 12-lead ECG was obtained in a semi-supine position after 5 minutes of rest at each indicated time point using an ECG machine that automatically calculated the heart rate and measured the PR, QRS, QT, and QT corrected by Fridericia's formula (QTcF) intervals. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: Baseline (Day -1) and Day 4 in each treatment period, and at Follow-up (at approximately Week 12)
Population: All Subjects
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | Placebo | Albiglutide 50 mg
Number analyzed (Participants) | 18 | 20
Milliseconds (msec)
  PR | 2.1 (8.58) | 2.2 (5.76)
  QRS | -1.8 (6.82) | -0.7 (4.46)
  QT | -5.0 (17.69) | -19.9 (21.08)
  QTcF | -7.7 (12.33) | -7.0 (15.85)

14. Secondary Outcome: Part A: Number of Participants With at Least One Non-serious Adverse Event (AE), Serious Adverse Event (SAE), or Drug-related Adverse Event
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, associated with liver injury and impaired liver function defined as alanine aminotransferase >=3 x upper limit of normal (ULN), and total bilirubin >=2 x ULN or international normalised ratio >1.5. AEs were classified as potentially drug-related, based on the investigator's judgement. Refer to the general AE/SAE module for a list of AEs and SAEs.
Time Frame: From Day -1 in treatment period 1 and up to Follow-up Visit (a total of approximately 12 weeks)
Population: All Subjects
Measure: Number; unit: Participants
Arm/Group | Placebo | Albiglutide 50 mg
Number analyzed (Participants) | 18 | 20
Participants
  Any AE | 8 | 9
  Any SAE | 0 | 0
  Any Drug-Related AE | 5 | 6

15. Secondary Outcome: Number of Participants for the Indicated Urinalysis Parameters Tested by Dipstick
Description: Urine dipstick test was carried out on Day -1 and at Follow-up. Urinalysis parameters assessed were glucose, ketones, nitrite and protein. Dipstick results were categorized as Normal (glucose), Negative or Trace (ketones), and Negative (nitrite and protein). Only participants available at the indicated time points (as represented by n=X, X, X in the category titles) were analyzed. The resultant fields with no available data have been represented by 'NA'.
Time Frame: Day -1 and Follow-up (assessed up to a total of approximately 12 weeks)
Population: All Subjects
Measure: Number; unit: Participants
Groups:
- Albiglutide 50 mg and Placebo: Participants were assessed at Follow-up after 28 days following the last dose of albiglutide or placebo.
Arm/Group | Placebo | Albiglutide 50 mg | Albiglutide 50 mg and Placebo
Number analyzed (Participants) | 18 | 20 | 20
Participants
  Urine Glucose Normal; Day -1; n=18, 20, 0 | 18 | 20 | NA — The result fields with no available data have be represented by NA.
  Urine Glucose Normal; Follow-up; n=0, 0, 19 | NA — The result fields with no available data have be represented by NA. | NA — The result fields with no available data have be represented by NA. | 19
  Urine Ketones Negative; Day -1; n=18, 20, 0 | 18 | 19 | NA — The result fields with no available data have be represented by NA.
  Urine Ketones Trace; Day -1; n=18, 20, 0 | 0 | 1 | NA — The result fields with no available data have be represented by NA.
  Urine Ketones Negative; Follow-up; n=0, 0, 19 | NA — The result fields with no available data have be represented by NA. | NA — The result fields with no available data have be represented by NA. | 19
  Urine Nitrite Negative; Day -1; n=18, 20, 0 | 18 | 20 | NA — The result fields with no available data have be represented by NA.
  Urine Nitrite Negative; Follow-up; n=0, 0, 19 | NA — The result fields with no available data have be represented by NA. | NA — The result fields with no available data have be represented by NA. | 19
  Urine Protein Negative; Day -1; n=17, 20, 0 | 17 | 20 | NA — The result fields with no available data have be represented by NA.
  Urine Protein Negative; Follow-up; n=0, 0, 18 | NA — The result fields with no available data have be represented by NA. | NA — The result fields with no available data have be represented by NA. | 18

ADVERSE EVENTS:
Time Frame: On-treament adverse events (AEs) and serious adverse events (SAEs) were collected from the start of study treatment and until the follow-up contact (a total of approximately 12 weeks)
Arm/Group | Placebo | Albiglutide 50 mg
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 8/18 | 9/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | Albiglutide 50 mg (N=20)
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dizziness postural (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Abdominal painv (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Feeling abnormal (General disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 1
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.